CLINICAL TRIAL: NCT01041092
Title: Double Blind, Placebo-controlled Study of Efficacy, Safety and Tolerance of Raloxifene as an Adjuvant Treatment for Negative Symptoms of Schizophrenia in Postmenopausal Women
Brief Title: Double Blind, Placebo-controlled Study of Raloxifene for Negative Symptoms of Schizophrenia in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Fundació Sant Joan de Deu
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04T-504
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator)
  Interventions: Drug: raloxifene
- raloxifene hydrochloride (Active Comparator): Dose of raloxifene hydrochloride will be: 60mg /day. Patients are required to continue taking their regular medications throughout the duration of the study. No changes in dose will be required during the study period. Double-blind treatment will continue for 12 weeks.
  Interventions: Drug: raloxifene

INTERVENTIONS:
Drug: raloxifene — Dose of raloxifene hydrochloride will be: 60mg /day. Patients are required to continue taking their regular medications throughout the duration of the study. No changes in dose will be required during the study period. Double-blind treatment will continue for 12 weeks.

SUMMARY:
Primary objective: To assess the efficacy of adding raloxifene as an adjunct to antipsychotic treatment to improve negative symptoms of schizophrenia in postmenopausal women.

This is a double-blind, randomized, placebo-controlled study of raloxifene as adjuvant treatment to antipsychotic treatment. Treatment period of 12 weeks.

The primary result obtained is that women treated with 60 mg of raloxifene compared to those treated with a placebo show greater improvement in psychotic symptoms. The investigators also found improved response in some aspects of social functioning and neuropsychological functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (DSM-IV criteria)
* Postmenopausal patients. Postmenopause is defined as after a period of one year of spontaneous amenorrhea and a serum follicle stimulating hormone (FSH) level > 20IU/L.
* Stable doses of their current antipsychotic medication for at least a month prior to study initiation.
* Presence of significant negative symptoms (defined as one or more negative symptom score greater than 4 in the PANSS scale) (Kay 1987)
* Patients have to give written informed consent to participate in the study.

Exclusion Criteria:

* Patients with a substance abuse/dependence diagnosis in the previous six months.
* Mental retardation.
* Endocrine abnormalities, acute or chronic liver disease, impaired kidney function.
* History of thromboembolism, breast cancer, abnormal uterine bleeding, history of cerebrovascular accident.
* Patients taking hormone replacement therapy.
* Patients taking mood stabilizer medication that cannot be discontinued.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy end-point will be the change in the score of the PANSS negative subscale from baseline to follow-up assessment.

SECONDARY OUTCOMES:
Patients social and neuropsychological functioning will be evaluated, comparing baseline ratings to end-point.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Sant Joan de Déu, Esplugues de Llobregat, Spain

REFERENCES:
- [Derived] Huerta-Ramos E, Iniesta R, Ochoa S, Cobo J, Miquel E, Roca M, Serrano-Blanco A, Teba F, Usall J. Effects of raloxifene on cognition in postmenopausal women with schizophrenia: a double-blind, randomized, placebo-controlled trial. Eur Neuropsychopharmacol. 2014 Feb;24(2):223-31. doi: 10.1016/j.euroneuro.2013.11.012. Epub 2013 Dec 1. PMID 24342775
- [Derived] Usall J, Huerta-Ramos E, Iniesta R, Cobo J, Araya S, Roca M, Serrano-Blanco A, Teba F, Ochoa S. Raloxifene as an adjunctive treatment for postmenopausal women with schizophrenia: a double-blind, randomized, placebo-controlled trial. J Clin Psychiatry. 2011 Nov;72(11):1552-7. doi: 10.4088/JCP.10m06610. Epub 2011 Aug 23. PMID 21903021